CLINICAL TRIAL: NCT04371068
Title: Evaluation of the microDTTect Device (Heraeus) in the Diagnosis of Low-grade Chronic
Brief Title: Heraeus MicroDTTect Lyon Pilot Studyprosthetic Joint Infections (PJIs)
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, clinical research assistant, Hospices Civils de Lyon
Other Study IDs: 18-265
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Chronic PJIs
Keywords: bone and joint infection; biofilm; joint arthroplasty; implant failure; prosthetic joint infection; dithiothreitol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suspected of low-grade PJIs: Adult patients suspected of low-grade PJIs, who have a scheduled prosthesis removal or change and who meet the inclusion criteria
  Interventions: Biological: Culture of removed prosthesis using DTT

INTERVENTIONS:
Biological: Culture of removed prosthesis using DTT — No specific or supplementary intervention is performed among patients. The included patients have scheduled surgery consisting of prosthesis removal or change. Instead of being discarded, the prosthesis which was removed during the surgery was sent to the laboratory using the MicroDTTect system and bacterial culture was performed with the fluid obtained. Results will be then compared to classical culture of periprosthetic tissues (PPT).

SUMMARY:
Prosthetic joint infections (PJIs) are one of the main causes of implant failure after joint arthroplasty. Identification of the causal organism is crucial for successful treatment. However, microbiological diagnosis of PJIs remains a challenge notably because bacteria are embedded in biofilm adhered to the material. Recently, dithiothreitol (DTT) treatment of prosthesis has been proposed as a new strategy to dislodge bacteria from biofilm, thus becoming an alternative to sonication to improve the yield of the microbiological diagnosis.

In this study, the investigators evaluate the interest of a commercial device using DTT, the MicroDTTect system (Heraeus, Hanau, Allemagne), for the diagnosis of low-grade chronic PJIs compared to the conventional culture of periprosthetic tissue (PPT) samples.

DETAILED DESCRIPTION:
Prosthetic joint infections (PJIs) are one of the main causes of implant failure after joint arthroplasty. Identification of the causal organism is crucial for successful treatment. However, microbiological diagnosis of PJIs remains a challenge notably because bacteria are embedded in biofilm adhered to the material. Recently, dithiothreitol (DTT) treatment of prosthesis has been proposed as a new strategy to dislodge bacteria from biofilm, thus becoming an alternative to sonication to improve the yield of the microbiological diagnosis.

In this study, the investigators evaluate the interest of a commercial device using DTT, the MicroDTTect system (Heraeus, Hanau, Allemagne), for the diagnosis of low-grade chronic PJIs compared to the conventional culture of periprosthetic tissue (PPT) samples.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with painful prosthesis or prosthesis loosening <10 years

* without mechanical explanation,
* without clinical evidence of infection (no fistula, no abscess, no discharge, no local inflammation),
* without microbiological diagnosis (absence of preoperative joint puncture (not performed or not feasible) or with a culture-negative preoperative joint puncture).

Exclusion Criteria:

Patients with painful prosthesis or prosthesis loosening

* with mechanical explanation,
* or with clinical evidence of infection (fistula, abscess, discharge, local inflammation),
* with a previous microbiological diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with painful prosthesis or prosthesis loosening <10 years treated at the CRIOAc Lyon
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of bacteria isolated isolated | every day until 15 days of culture
  type of bacteria isolated

SECONDARY OUTCOMES:
time to positivity of cultures | every day until 15 days of culture
  time to positivity of cultures of the fluid obtained after prosthesis treatment using the MicroDTTect system in comparison with conventional culture of PPT samples

CONTACTS AND LOCATIONS:
Overall Officials: FREDERIC LAURENT, Principal Investigator — LAURENT
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: website of CRIOAc Lyon — http://www.crioac-lyon.fr